CLINICAL TRIAL: NCT05643703
Title: A Prospective Randomized Controlled Study on the Efficacy and Safety of Different Suture Methods for the Transvaginal Repair of Cesarean Section Defect and the Exploration of the Underlying Molecular Mechanism of the Defect Occurrence
Brief Title: Cesarean Section Defect Mechanism and Transvaginal Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K2724
Record Dates: First submitted 2022-11-29; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Cesarean Scar Defect; Transvaginal Diverticulum Resection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-layered Suture (Experimental): One-layered Suture in transvaginal diverticulum resection
  Interventions: Procedure: Suture method
- Two-layered Suture (Experimental): Two-layered Suture in transvaginal diverticulum resection
  Interventions: Procedure: Suture method

INTERVENTIONS:
Procedure: Suture method — One-layered Suture: Single layer intermittent suture; Two-layered Suture:Single layer intermittent suture plus U type reinforcement stitching

SUMMARY:
Background and aims: Cesarean section defect (CSD) can cause abnormal uterine bleeding or impaired fertility, which severely impaire the quality of life in women of pregnant age. For women with moderate or severe CSD, surgery can be performed. The objectives of this study is to compare the efficacy and safety of different suture methods in the treatment of transvaginal diverticulum resection, and the underlying mechanism of CSD occurrence.

Methods: The patients diagnosed with CSD will be enrolled and randomizely assigned into suture method A and suture method. The fresh isolated tissue and swab of different sites in genital tract will be collected for NGS, microbiome, metabonomics and proteomics analysis.

Hypothesis: The menstruation will be analyzed at different following time. The other clinical information will be also collected, including age at surgery, skin-to skin operative time, estimated blood loss (EBL). The perioperative complications, postoperative hopitalization, cost for hospital stay, blasser/intestinal function recovery will also be compared between two gorup. The outcome of fertility will be compared, such as the premature birth, premature rupture of membranes, and rupture of uterus. The clinical manifestation related to CSD and recurrence will be followed. Besides, the underlying mechanism will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, premenopausal female;
2. The scar is the transverse incision of the lower segment of the uterus (one or more times);
3. The following abnormal uterine bleeding occurred after cesarean section: prolonged menstruation/endless menstruation ≥ 14 days, menstrual bleeding;
4. Transvaginal three-dimensional ultrasound/pelvic MRI plain scan showed that the thickness of residual muscular layer at the top of diverticulum was less than 3 mm;
5. The effect of drug treatment is poor, and it is difficult to adhere to long-term drug treatment or surgical treatment;
6. HGB > 100g/L before operation;
7. Hysteroscopy excluded endometrial lesions;
8. The patient or family members can understand the study protocol and voluntarily participate in the study, and provide written informed consent.

Exclusion Criteria:

1. The data of cesarean section is not complete, and the previous cesarean section method cannot be determined;
2. Abnormal uterine bleeding caused by endocrine disorders (thyroid dysfunction, luteal insufficiency), endometrial lesions, uterine fibroids, gynecological tumors, blood system diseases, pelvic infections, intrauterine devices, etc;
3. Infertility patients caused by female oviduct infertility, intrauterine adhesion infertility, uterine malformation, polycystic ovary syndrome, male infertility, etc;
4. Patients with other serious gynecological diseases and/or serious physical or psychological diseases;
5. Pregnancy (women of childbearing age were positive in pregnancy test at baseline or did not receive pregnancy test), and women in lactation;
6. Patients who are unable to complete the follow-up;
7. The patient or family members could not understand the conditions and objectives of the study and did not agree to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Prolongation of menstrual period | 3 month after surgery
  Patients' subject description of the duration of menstrual period, which is defined as the first day of menstruation to the end day

SECONDARY OUTCOMES:
fertility outcome | within 5 years after surgery
  record the post-operative fertility outcome, including natural pregnancy or assisted reproduction, and the correspondence fertility outcome, such as premature birth, premature rupture of membranes, etc.

OTHER OUTCOMES:
objective measurement of caesarean scar diverticulum | within 1 years after surgery
  The difference of different diameters of caesarean scar diverticulum before and after surgery